CLINICAL TRIAL: NCT00216775
Title: Comparative Trial of Standard Versus Low-dose Peg-Interferon Plus Ribavirin in the Treatment of Chronic Hepatitis C
Status: Completed | Type: Observational
Sponsor: Kyoto University (Other)
Responsible Party: Principal Investigator, Hiroyuki Marusawa, Dep Gastroenterol, Kyoto University
Organization: Kyoto University Hospital (Other)
Other Study IDs: H16-697
Record Dates: First submitted 2005-09-10; First posted 2005-09-22 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-09

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Introns; Ribavirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Drug: interferon-alfa-2b and ribavirin

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of low-dose interferon-alfa-2b plus ribavirin compared to the standard-dose of the same combination in patients with chronic hepatitis C.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Chronic Hepatitis C. Must be infected with genotype 1b viruses

Exclusion Criteria:

* Hemoglobin levels<8.5g/dL,
* Platelet counts<50,000/mm3,
* Total polymorphonuclear counts<1000/mm3
* Pregnancy,
* Renal dysfunction,

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with chronic hepatitis C
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2004-12; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
rate of sustained viral response | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Tsutomu Chiba, M.D., Ph.D, Study Chair — Kyoto University Hospital
Locations (4):
- Japan (4):
  - Department of Gastroenterology and Hepatology, Kyoto University Hospital, Kyoto
  - Kitano Hospital, Osaka
  - Osaka Red Cross Hospital, Osaka
  - Wakayama Red Cross Hospital, Wakayama